CLINICAL TRIAL: NCT06227078
Title: Clinical and Functional Effects of Kinesiotaping and Physiotherapy in Grade 2 Osteoarthritis Following Degenerative Meniscal Tears in Football Players - A Randomized Control Trial
Brief Title: Effects of Kinesiotaping and Physiotherapy in Grade 2 Osteoarthritis Following Degenerative Meniscal Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gopal Nambi (Other)
Responsible Party: Sponsor-Investigator, Gopal Nambi, Gopal Nambi, Prince Sattam Bin Abdulaziz University
Organization: Prince Sattam Bin Abdulaziz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/021/093
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis; Meniscus Tear
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Kinesiotaping + Physiotherapy (Active Comparator): The application of kinesiotaping for grade 2 osteoarthritis involves the application of an anchor strip at one end of the affected joint, typically with no stretch. Apply the kinesiotape with the desired amount of stretch, usually around 50-80% of its maximum stretch capacity. Direct the tape along the muscle or joint in a specific pattern, such as "I," "Y," or "X" depending on the therapeutic goal. Finish with an anchor strip at the opposite end, with no stretch to secure the tape in place.
  Physiotherapy:
  Apply TENS: Low-frequency TENS (2-10 Hz) that produces a tingling or buzzing sensation without causing discomfort or pain. TENS sessions may last between 20 to 30 minutes per session.
  Strengthening exercises:
  1. Quadriceps Sets:
  2. Straight Leg Raises:
  3. Seated Leg Press:
  4. Hamstring Curls:
  5. Calf Raises:
     * Repeat the exercises for 10 times, 3 sets in a session for 8 weeks.
  Interventions: Device: Kinesiotaping
- Placebo Kinesiotaping + Physiotherapy (Placebo Comparator): The application of kinesiotaping for grade 2 osteoarthritis involves the application of an anchor strip at one end of the affected joint, typically with no stretch. Apply the kinesiotape without stretch, Direct the tape along the muscle or joint in a specific pattern, such as "I," "Y," or "X" depending on the therapeutic goal. Finish with an anchor strip at the opposite end, with no stretch to secure the tape in place.
  Physiotherapy:
  Apply TENS: Low-frequency TENS (2-10 Hz) that produces a tingling or buzzing sensation without causing discomfort or pain. TENS sessions may last between 20 to 30 minutes per session.
  Strengthening exercises:
  1. Quadriceps Sets:
  2. Straight Leg Raises:
  3. Seated Leg Press:
  4. Hamstring Curls:
  5. Calf Raises:
     * Repeat the exercises for 10 times, 3 sets in a session for 8 weeks.
  Interventions: Device: Kinesiotaping

INTERVENTIONS:
Device: Kinesiotaping — Kinesiotaping is commonly used in sports medicine and rehabilitation settings. It is applied by trained professionals, such as physiotherapists or athletic trainers, who are skilled in assessing individual needs and determining the appropriate taping technique for specific conditions. The tape is typically worn for several days, allowing for continuous therapeutic effects.
  It's important to note that while kinesiotaping has gained popularity, its effectiveness is still a subject of ongoing research, and its application should be part of a comprehensive treatment plan. Individual responses to kinesiotape may vary, and its use is often combined with other therapeutic interventions for optimal results.

SUMMARY:
Degenerative meniscal tears are a common cause of osteoarthritis commonly diagnosed in football players and are considered a major risk factor for the development of knee osteoarthritis. This study aimed to investigate the Clinical and functional effects of kinesiotaping and physiotherapy in grade 2 osteoarthritis following degenerative meniscal tears in football players.

DETAILED DESCRIPTION:
Degenerative meniscal tears represent a prevalent issue among football players and are frequently associated with an increased risk of developing knee osteoarthritis. This study seeks to explore the clinical and functional impacts of employing kinesiotaping and physiotherapy as interventions in grade 2 osteoarthritis resulting from degenerative meniscal tears in football players.

Kinesiotaping is a therapeutic technique involving the application of specialized elastic tapes to targeted areas, aiming to support injured muscles and joints, enhance circulation, and alleviate pain. Physiotherapy, on the other hand, employs a range of exercises and modalities to promote healing and improve joint function. Both modalities are commonly used in sports medicine to manage musculoskeletal injuries.

The investigation focuses on football players diagnosed with grade 2 osteoarthritis secondary to degenerative meniscal tears. Grade 2 osteoarthritis signifies moderate cartilage loss and potential joint instability. The participants will be divided into two groups: one receiving kinesiotaping in combination with physiotherapy and the other undergoing conventional physiotherapy alone.

Clinical assessments will include pain levels, joint swelling, and range of motion. Functional outcomes such as strength, agility, and proprioception will be measured through standardized tests. The study's duration and follow-up periods will allow for a comprehensive evaluation of both short-term and long-term effects.

The hypothesis underlying this research posits that the combined approach of kinesiotaping and physiotherapy will yield superior outcomes compared to traditional physiotherapy alone. Potential benefits may include reduced pain, improved joint stability, enhanced functional capacity, and a decreased risk of further degeneration.

By shedding light on the efficacy of these interventions, this study aspires to contribute valuable insights to the field of sports medicine, aiding in the development of evidence-based strategies for managing degenerative meniscal tears and mitigating the risk of osteoarthritis in football players. The findings could inform clinical practice and potentially influence rehabilitation protocols for athletes facing similar challenges.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Knee Osteoarthritis:

Individuals with a confirmed diagnosis of knee osteoarthritis based on clinical and/or radiological assessments.

Mild to Moderate Knee OA:

Kinesiotaping may be more appropriate for individuals with mild to moderate knee OA rather than severe cases.

Presence of Pain and Discomfort:

Individuals experiencing pain, discomfort, or limitations in function related to knee osteoarthritis.

Functional Limitations:

Those with functional limitations in activities of daily living or reduced mobility due to knee OA.

No Contraindications:

Individuals without contraindications to kinesiotaping, such as skin allergies, infections, or open wounds in the application area.

Willingness to Participate:

Individuals who are willing to participate in and adhere to the kinesiotaping intervention.

Not Responsive to Other Conservative Treatments:

Those who have tried and not responded adequately to other conservative treatments for knee OA, such as exercise, physical therapy, or oral medications.

Absence of Serious Comorbidities:

Individuals without serious comorbidities or medical conditions that may contraindicate the use of kinesiotaping.

Individual Preferences:

Consideration of individual preferences and acceptance of kinesiotaping as part of the treatment plan.

Exclusion Criteria:

* 1. Skin Conditions:

  * Active skin infections, allergies, or open wounds in the area where kinesiotape is to be applied.
  * Skin conditions that may be aggravated or worsened by the adhesive in the tape. 2. Vascular Disorders:
  * Conditions that affect blood circulation, such as peripheral vascular disease, deep vein thrombosis, or other vascular disorders, which may be worsened by the application of kinesiotape.

    3. Peripheral Neuropathy:
  * Individuals with peripheral neuropathy or other nerve disorders, as kinesiotaping may affect sensation, and there is a risk of injury or discomfort.

    4. Cancer or Tumors:
  * Active cancer or tumors in the region where kinesiotape is to be applied, as kinesiotaping could interfere with cancer treatment or exacerbate symptoms.

    5. Joint Instability:
  * Individuals with severe joint instability, as kinesiotape may not provide sufficient support for highly unstable joints.

    6. Allergies to Tape Components:
  * Known allergies to the materials or adhesive used in kinesiotape. 7. Circulatory Disorders:
  * Severe circulatory disorders, which may be exacerbated by the pressure or tension applied by kinesiotape.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity - Visual analog scale | Baseline
  The VAS is usually presented as a straight line, often 10 centimeters (or another standard length), with two endpoints representing extreme points on a continuum. For example, one end may be labeled "No Pain" or "No Symptoms," and the other end labeled "Worst Pain Imaginable" or "Maximum Symptoms."
Pain intensity - Visual analog scale | 8 weeks
  The VAS is usually presented as a straight line, often 10 centimeters (or another standard length), with two endpoints representing extreme points on a continuum. For example, one end may be labeled "No Pain" or "No Symptoms," and the other end labeled "Worst Pain Imaginable" or "Maximum Symptoms."
Pain intensity - Visual analog scale | 6 months
  The VAS is usually presented as a straight line, often 10 centimeters (or another standard length), with two endpoints representing extreme points on a continuum. For example, one end may be labeled "No Pain" or "No Symptoms," and the other end labeled "Worst Pain Imaginable" or "Maximum Symptoms."

SECONDARY OUTCOMES:
Functional disability - WOMAC | Baseline
  The WOMAC scale consists of three subscales, each assessing a different dimension of health related to osteoarthritis.
Functional disability - WOMAC | 8 weeks
  The WOMAC scale consists of three subscales, each assessing a different dimension of health related to osteoarthritis.
Functional disability - WOMAC | 6 months
  The WOMAC scale consists of three subscales, each assessing a different dimension of health related to osteoarthritis.
Sports performance - Timed up and go test | Baseline
  Ask the individual to sit in the chair with their back against the backrest and their arms on the chair arms (if available). On the "go" signal, instruct them to stand up, walk around the first cone, return to the chair, and sit back down. Use a stopwatch to measure the time it takes for the individual to complete the task. Faster times generally indicate better agility and functional mobility.
Sports performance - Timed up and go test | 8 weeks
  Ask the individual to sit in the chair with their back against the backrest and their arms on the chair arms (if available). On the "go" signal, instruct them to stand up, walk around the first cone, return to the chair, and sit back down. Use a stopwatch to measure the time it takes for the individual to complete the task. Faster times generally indicate better agility and functional mobility.
Sports performance - Timed up and go test | 6 months
  Ask the individual to sit in the chair with their back against the backrest and their arms on the chair arms (if available). On the "go" signal, instruct them to stand up, walk around the first cone, return to the chair, and sit back down. Use a stopwatch to measure the time it takes for the individual to complete the task. Faster times generally indicate better agility and functional mobility.
Sports performance - 40 Metre zig zag test | Baseline
  Set up a zigzagging path using cones or markers. The path should be 40 meters in total length. The zigzag pattern should include sharp turns, requiring participants to change direction quickly. Explain the test to the participant, emphasizing the need to navigate through the zigzag path as quickly as possible.
  Emphasize the importance of agility, speed, and quick changes in direction. Use a stopwatch or timer to measure the time it takes for the participant to complete the 40-meter zigzag course. On the "go" signal, the participant should start from the beginning and navigate through the zigzag path as quickly as possible.
  Time should be recorded when the participant crosses the finishing line.
Sports performance - 40 Metre zig zag test | 8 weeks
  Set up a zigzagging path using cones or markers. The path should be 40 meters in total length. The zigzag pattern should include sharp turns, requiring participants to change direction quickly. Explain the test to the participant, emphasizing the need to navigate through the zigzag path as quickly as possible.
  Emphasize the importance of agility, speed, and quick changes in direction. Use a stopwatch or timer to measure the time it takes for the participant to complete the 40-meter zigzag course. On the "go" signal, the participant should start from the beginning and navigate through the zigzag path as quickly as possible.
  Time should be recorded when the participant crosses the finishing line.
Sports performance - 40 Metre zig zag test | 6 months
  Set up a zigzagging path using cones or markers. The path should be 40 meters in total length. The zigzag pattern should include sharp turns, requiring participants to change direction quickly. Explain the test to the participant, emphasizing the need to navigate through the zigzag path as quickly as possible.
  Emphasize the importance of agility, speed, and quick changes in direction. Use a stopwatch or timer to measure the time it takes for the participant to complete the 40-meter zigzag course. On the "go" signal, the participant should start from the beginning and navigate through the zigzag path as quickly as possible.
  Time should be recorded when the participant crosses the finishing line.
Quality of life - SF-12 | Baseline
  The Short Form Health Survey (SF-12) is a widely used and validated questionnaire designed to assess health-related quality of life (HRQoL) across various populations. It is a shorter version of the SF-36 and provides a quick and reliable measure of general health status. The SF-12 includes 12 questions covering eight health domains and yields two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
Quality of life - SF-12 | 8 weeks
  The Short Form Health Survey (SF-12) is a widely used and validated questionnaire designed to assess health-related quality of life (HRQoL) across various populations. It is a shorter version of the SF-36 and provides a quick and reliable measure of general health status. The SF-12 includes 12 questions covering eight health domains and yields two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
Quality of life - SF-12 | 6 months
  The Short Form Health Survey (SF-12) is a widely used and validated questionnaire designed to assess health-related quality of life (HRQoL) across various populations. It is a shorter version of the SF-36 and provides a quick and reliable measure of general health status. The SF-12 includes 12 questions covering eight health domains and yields two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).

CONTACTS AND LOCATIONS:
Locations (1):
- Saud Alrawilli, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: 2 months